CLINICAL TRIAL: NCT06453408
Title: Validation of a Placebo Dry Needling Protocol in Patients With Non-specific Neck Pain: a Randomised Controlled Clinical Trial
Brief Title: Validation of a Placebo Dry Needling Protocol in Patients With Non-specific Neck Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Leire Vázquez Casar, Leire Vázquez Casar, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PS-Leire
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Neck Pain
Keywords: dry needling; validation; placebo; neck pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo, sin experiencia (Sham Comparator): Group of patients with no previous experience in dry needling, will be given placebo dry needling
  Interventions: Procedure: Punción seca con aguja retráctil
- Placebo, con experiencia (Sham Comparator): Group of patients with previous experience in dry needling, will be given placebo dry needling
  Interventions: Procedure: Punción seca con aguja retráctil
- Real, sin experiencia (Experimental): Group of patients with no previous experience in dry needling, real dry needling will be applied
  Interventions: Procedure: Punción seca con aguja normativa.
- Real, con experiencia (Experimental): Group of patients with previous experience in dry needling, real dry needling will be applied.
  Interventions: Procedure: Punción seca con aguja normativa.

INTERVENTIONS:
Procedure: Punción seca con aguja retráctil — The placebo dry needling protocol will be performed in the same position, with identical antiseptic measures and the same number of simulated incisions as the real dry needling protocol, using DONGBANG AcuPrime® 0.30 x 30mm blunt-tipped placebo needles with a retractable handle. These needles simulate the sensation of needle contact without penetrating the skin. The therapist will hold the needle and guide tube, pressing the tube against the skin and simulating needle manipulation. Changes in pressure direction will mimic the real technique. The protocol will end with compression using an alcohol swab and an upper trapezius stretch.
  Participants in both groups will receive the same information about the sensations of the dry needling procedure. At the beginning, they will be informed that they may or may not feel the needle insertion. They will also be told that the physiotherapist will manually manipulate the needle multiple times during the procedure.
  Other Names: DONGBANG AcuPrime® de 0,30 x 30mm.
  Arms: Placebo, con experiencia; Placebo, sin experiencia
Procedure: Punción seca con aguja normativa. — To perform the actual SP, patients shall be asked to lie prone with arms close to the body. The dry needling shall be performed with a 0,30 × 30 mm DN needle (APS Regular Agupunt) with a guide tube. The therapist shall first clean the area with alcohol. The trapezius muscle is then firmly grasped with a clamp between the thumb and index finger, so that the needle is directed deep into the index finger until the tip of the needle is felt to be approaching (33). This procedure involves an approximate insertion of the needle to a depth of 30 mm and ensures the intramuscular penetration necessary for dry needling. Puncture of the PGM shall be performed using the Hong technique (34), performing up to 12 inlets and outlets, at a frequency of 1 Hz. When the needle is withdrawn, the area is firmly compressed with cotton wool for 60 seconds. Finally, the upper trapezius muscle is stretched, following the technique originally described by Simons (35).
  Other Names: APS Regular Agupunt 0,30 × 30 mm
  Arms: Real, con experiencia; Real, sin experiencia

SUMMARY:
This study aims to validate a placebo dry needling protocol for patients with non-specific neck pain and investigate whether prior experience with dry needling affects their ability to distinguish between real and placebo treatments, and how this impacts outcomes. Seventy participants aged 18-65 will be recruited and divided into two groups based on their previous dry needling experience, then randomized into real or placebo needling groups.

Assessment will be carried out before treatment, immediately after the procedure and one week later. Pain intensity, pain threshold to pressure, cervical range of motion, level of disability and presence of central sensitisation will also be measured.

DETAILED DESCRIPTION:
Background: There is currently no valid and reliable method available to perform a placebo dry needling protocol in patients with non-specific neck pain. The lack of uniformity and validity in placebo dry needling methods hinders research on the specific effects of this technique. In addition, there is no solid evidence on how patients' previous experiences affect their expectations of treatment. An effective placebo dry needling protocol is essential for future research on the effectiveness of dry needling in randomised controlled clinical trials.

Objective: The main objective of this study is to validate a placebo dry needling protocol. The secondary objective is to examine whether the patient's previous experience with dry needling influences their ability to discern between having received a real or placebo needling and how this impacts on the outcomes of the intervention.

Material and method: 70 participants aged 18-65 years with non-specific neck pain who meet the inclusion criteria will be recruited. They will be assigned to one of two groups, those who have previously received dry needling and those who have not. Thereafter, members of each group will be randomised and assigned to either the real dry needling or placebo group. Assessment will be carried out before treatment, immediately after the procedure and one week later. Pain intensity, pain threshold to pressure, cervical range of motion, level of disability and presence of central sensitisation will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific neck pain, unilateral or bilateral.
* Neck pain lasting ≥ 3 months.
* Presence of active myofascial trigger point (MTrP) in the upper trapezius muscle, left, right or bilateral, in relation to the patient's neck pain.

Exclusion Criteria:

* Fear or phobia of needles
* Skin lesions, infection or inflammation in the area to be pricked
* Specific alterations of the cervical region in the medical history
* Coagulation disorders
* Surgical intervention of the cervical or anterior shoulder region
* Undergoing pharmacological treatment with analgesics, anti-inflammatory drugs or anticoagulants in the week prior to the study.
* Having received physiotherapy treatment in the neck region in the 6 months prior to the intervention.
* Infiltration of corticosteroids or local anaesthetics up to one year prior to the study.
* Cognitive deficits in the medical history.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-06-25 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Successful identification rate of group assignment | Immediately after the intervention and one week later, in order to see if any participants change their response.
  A Questionnaire of its own, designed to record participants' perceptions of the perceived intervention, will be used. Participants will be asked to select which group they believe they belong to by choosing one of five possible responses:
  1. I strongly believe I was assigned to the treatment group.
  2. I believe to some extent that I was assigned to the treatment group.
  3. I believe to some extent that I was assigned to the control group.
  4. I strongly believe that I was assigned to the control group.
  5. I am not sure

SECONDARY OUTCOMES:
Pain intensity | Before and immediately after the intervention, and a new assessment will be carried out one week later.
  Visual Analogic Scale
Neck disability | Before and one week after the intervention.
  neck disability index
Cervical Range of Motion | Before intervention, immediately after intervention and after one week.
  Grades
central sensitisation | Before the intervention and one week after
  The Central Sensitisation Inventory (CSI)
Pressure pain threshold | Before the intervention, immediately after the intervention and one week afterwards
  kg/sec

CONTACTS AND LOCATIONS:
Overall Officials: Leire Vazquez-Casar, Principal Investigator — University of Alcala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pariente J, White P, Frackowiak RS, Lewith G. Expectancy and belief modulate the neuronal substrates of pain treated by acupuncture. Neuroimage. 2005 May 1;25(4):1161-7. doi: 10.1016/j.neuroimage.2005.01.016. PMID 15850733
- [Background] Bier JD, Scholten-Peeters WGM, Staal JB, Pool J, van Tulder MW, Beekman E, Knoop J, Meerhoff G, Verhagen AP. Clinical Practice Guideline for Physical Therapy Assessment and Treatment in Patients With Nonspecific Neck Pain. Phys Ther. 2018 Mar 1;98(3):162-171. doi: 10.1093/ptj/pzx118. PMID 29228289
- [Background] Boonstra AM, Schiphorst Preuper HR, Reneman MF, Posthumus JB, Stewart RE. Reliability and validity of the visual analogue scale for disability in patients with chronic musculoskeletal pain. Int J Rehabil Res. 2008 Jun;31(2):165-9. doi: 10.1097/MRR.0b013e3282fc0f93. PMID 18467932
- [Background] Andrade Ortega JA, Delgado Martinez AD, Almecija Ruiz R. [Validation of a Spanish version of the Neck Disability Index]. Med Clin (Barc). 2008 Feb 2;130(3):85-9. doi: 10.1157/13115352. Spanish. PMID 18261377
- [Background] Cuesta-Vargas AI, Roldan-Jimenez C, Neblett R, Gatchel RJ. Cross-cultural adaptation and validity of the Spanish central sensitization inventory. Springerplus. 2016 Oct 21;5(1):1837. doi: 10.1186/s40064-016-3515-4. eCollection 2016. PMID 27818875
- [Background] Baldry P. Superficial versus deep dry needling. Acupunct Med. 2002 Aug;20(2-3):78-81. doi: 10.1136/aim.20.2-3.78. PMID 12216605
- [Background] Hafliethadottir SH, Juhl CB, Nielsen SM, Henriksen M, Harris IA, Bliddal H, Christensen R. Placebo response and effect in randomized clinical trials: meta-research with focus on contextual effects. Trials. 2021 Jul 26;22(1):493. doi: 10.1186/s13063-021-05454-8. PMID 34311793
- [Background] Birch S. A review and analysis of placebo treatments, placebo effects, and placebo controls in trials of medical procedures when sham is not inert. J Altern Complement Med. 2006 Apr;12(3):303-10. doi: 10.1089/acm.2006.12.303. PMID 16646730
- [Background] Bang H, Ni L, Davis CE. Assessment of blinding in clinical trials. Control Clin Trials. 2004 Apr;25(2):143-56. doi: 10.1016/j.cct.2003.10.016. PMID 15020033
- [Background] Rodriguez-Huguet M, Vinolo-Gil MJ, Gongora-Rodriguez J. Dry Needling in Physical Therapy Treatment of Chronic Neck Pain: Systematic Review. J Clin Med. 2022 Apr 23;11(9):2370. doi: 10.3390/jcm11092370. PMID 35566496